CLINICAL TRIAL: NCT01848730
Title: A Randomised Double-blind Crossover Study to Compare the Efficacy and Safety of CNV2197944 75 mg Tid Versus Placebo in Patients With Post-herpetic Neuralgia
Brief Title: Efficacy and Safety of CNV2197944 Versus Placebo in Patients With Post-herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Convergence Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNV2197944/201
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-01

CONDITIONS: Post-herpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNV2197944 (Experimental): CNV2197944 75mg tid 21 days
  Interventions: Drug: CNV2197944
- Placebo (Placebo Comparator): Placebo tid 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNV2197944
  Arms: CNV2197944
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the effect of repeat oral dosing of CNV2197944 75 mg tid on the pain experienced in post-herpetic neuralgia (PHN) as measured by changes in PI-NRS after three weeks of treatment compared to the baseline period.

DETAILED DESCRIPTION:
A 3 week randomised crossover study to investigate the effect of repeat oral dosing of CNV2197944 75 mg tid versus placebo for on the pain experienced in post-herpetic neuralgia (PHN. Each 3 week treatment period is seperated by a 2 week washout period. The primary outcome measure is the change from baseline in the PI-NRS after three weeks of treatment. Secondary outcome measures include pain responder rates, clinical and patient global impressions of pain, and the Neuropathic Pain Symptom Inventory.

ELIGIBILITY:
Inclusion Criteria:

Male or female between 18 and 85 years of age inclusive, at the time of signing the informed consent.

Patients with post-herpetic neuralgia (PHN) with pain at screening present for more than 3 months after healing of the herpes zoster skin rash. The maximum duration of PHN will be no longer than 5 years.

Exclusion Criteria:

Patients having other severe pain, which may impair the self-assessment of the pain due to PHN.

Patients who have received nerve blocks for neuropathic pain within 4 weeks prior to the start of the single-blind placebo run-in Certain medications used to relieve the pain of PHN, specifically gabapentinoids (gabapentin and pregabalin), carbamazepine and topical agents (eg capsaicin, lidocaine) Patients with a documented failure to respond to a maximally tolerated dose regimen of gabapentin or pregabalin.

Patients taking more than one medication to treat the PHN pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Numerical Rating Scale | 21 days

SECONDARY OUTCOMES:
Pain responder rates | 21 days
Neuropathic Pain Symptom Inventory | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Milton Raff, MD, Principal Investigator — Christiaan Barnard Memorial Hospital, Cape Town, South Africa
Locations (1):
- Christiaan Barnard Memorial Hospital, Cape Town, South Africa